CLINICAL TRIAL: NCT04893889
Title: Substudy (NCT04456582): Noninvasive Assessment of Myocardial Stiffness by 2D-SWE Ultrasound Technique (Two-dimensional Shear Wave Elastography) in Patients With Amyloidosis and Fabry Disease.
Acronym: FABRY
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Sao Paulo General Hospital (Other)
Collaborators: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Diagnostic
Other Study IDs: 4963/19/182 FABRY
Record Dates: First submitted 2021-05-14; First posted 2021-05-20 (Actual); Last update posted 2021-05-20 (Actual); Status verified 2021-04

CONDITIONS: Fabry Disease; Amyloidosis
Keywords: Fabry disease; Amyloidosis; Shear-wave elastography
MeSH Terms: conditions — Fabry Disease; Amyloidosis

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Fabry disease patients (Experimental): Patients diagnosed with Fabry disease. Interventions will be as follows: Shear wave myocardial elastography to assess myocardial stiffness by non-invasively quantifying diastolic myocardial elasticity (EMD) in Fabry disease (DF) and cardiac amyloidosis (AC) in the ATTRh form and correlating with other complementary imaging tests and laboratory tests (electrocardiogram, 2D echocardiogram, troponin and BNP) and with a 6-minute walk test and quality of life questionnaires.
  Interventions: Diagnostic Test: Shear-wave elastography
- Amyloidosis transthyretin with cardiac commitment (Active Comparator): Patients diagnosed with amyloidosis who present cardiac commitment. Interventions will be as follows: Shear wave myocardial elastography to assess myocardial stiffness by non-invasively quantifying diastolic myocardial elasticity (EMD) in Fabry disease (DF) and cardiac amyloidosis (AC) in the ATTRh form and correlating with other complementary imaging tests and laboratory tests (electrocardiogram, 2D echocardiogram, troponin and BNP) and with a 6-minute walk test and quality of life questionnaires.
  Interventions: Diagnostic Test: Shear-wave elastography
- Healthy subjects (Placebo Comparator): Healthy patients. Interventions will be as follows: Shear wave myocardial elastography to assess myocardial stiffness by non-invasively quantifying diastolic myocardial elasticity (EMD) in Fabry disease (DF) and cardiac amyloidosis (AC) in the ATTRh form and correlating with other complementary imaging tests and laboratory tests (electrocardiogram, 2D echocardiogram, troponin and BNP) and with a 6-minute walk test.
  Interventions: Diagnostic Test: Shear-wave elastography

INTERVENTIONS:
Diagnostic Test: Shear-wave elastography — Myocardial shear wave elastography to assess myocardial stiffness by non-invasively quantifying diastolic myocardial elasticity.

SUMMARY:
Introduction: Heart failure with preserved systolic function encompasses several different diseases, but which have diastolic dysfunction and its components in common: myocardial stiffness and altered relaxation. Myocardial stiffness represents an important parameter for diagnosis and prognosis, but only changes in relaxation are evaluated in clinical practice. Cardiac elastography has been proposed as a diagnostic modality for noninvasive assessment of myocardial stiffness.

Objective: The aim of our study is to investigate the potential of myocardial elastography by shear waves to assess myocardial stiffness by non-invasively quantifying diastolic myocardial elasticity (EMD) in Fabry disease (DF) and cardiac amyloidosis (AC ) in the ATTRh form and correlate with other complementary imaging and laboratory tests (electrocardiogram, 2D echocardiogram, troponin and BNP) and with a 6-minute walk test and quality of life questionnaires.

Material and methods: 60 adults will be prospectively included: 20 patients with Fabry disease, 40 patients with hRTRT (20 with cardiac involvement) and 20 patients as a control group. Echocardiography, electrocardiogram and laboratory evaluations will be performed. The elastocardiographic assessment of myocardial stiffness will be performed in ultrasound equipment (Canon, Aplio i800) using a multifrequency convex transducer, under specific adjustment of the equipment to perform myocardial elastography.

ELIGIBILITY:
Inclusion Criteria:

- Documented diagnosis of ATTRh with and without cardiac involvement.

For the definition of cardiac involvement by ATTRh, all the criteria below must be presented:

* Pathogenic mutation of TTR consistent with ATTRh.
* Evidence of cardiac commitment by echocardiography or nuclear magnetic resonance with measurement of the interventricular septum at the end of diastole (SIVd)> 12mm or / and medical history of heart failure, and / or levels of troponin and / or BNP above the reference value without another more likely cause.
* Amyloid deposit in cardiac or extra-cardiac tissue (eg, abdominal fat aspirate, salivary gland, connective sheath of the median nerve) confirmed by congo red staining or presence of grade 2 or 3 myocardial scintigraphy (DPD-CT) of cardiac uptake, in cases where the presence of monoclonal gammopathy of undetermined significance (MGUS) was ruled out.
* In the presence of MGUS, confirmation of the TTR protein in the tissue is necessary through immunohistochemistry (IHC) or mass spectrometry.

Exclusion Criteria:

* Presence of another type of cardiomyopathy such as hypertension, valve or ischemic heart disease (eg, previous myocardial infarction documented with myocardial necrosis markers and electrocardiographic changes).
* Presence of diseases other than cardiac amyloidosis, impairing the assessment of functional capacity, such as chronic obstructive pulmonary disease, severe arthritis or peripheral arterial disease, recent or planned orthopedic procedure during the course of the study (eg, spine surgery or under lower limbs) that impairs walking in the 6-minute test evaluation.
* Acute coronary heart disease or unstable angina in the past 3 months Report of disease of the sinus or atrioventricular node with indication of a pacemaker, but with no intention of implantation.
* Presence of untreated hypothyroidism or hyperthyroidism.
* Previous heart, liver or other organ transplant.
* Presence of neoplasia in the last 3 years, except for basal and squamous cell carcinomas of skin or cervical cancer in situ previously treated.
* Presence of other medical conditions or comorbidities that, in the investigator's opinion, could interfere with the course of the study or the interpretation of the data.
* Pregnancy.
* History of alcohol abuse in the last 2 years or excessive daily alcohol intake (for women, more than 14 units per week; for men, more than 21 units of alcohol per week [unit: one glass of wine (125ml) = one dose of distillate = 332.5ml of beer).

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2020-09-09 (Actual); Primary Completion 2021-08-31 (Estimated); Study Completion 2022-03-30 (Estimated)

PRIMARY OUTCOMES:
Myocardial stiffness | 7 months
  To evaluate the diastolic myocardial elasticity in patients with Fabry's disease and compare it with the ATTR group with cardiac involvement and the control group.

SECONDARY OUTCOMES:
Systolic and diastolic function | 7 months
  To correlate diastolic myocardial elasticity with systolic and diastolic function indexes assessed by two-dimensional echocardiogram and with strain analysis using the speckle tracking technique;
Brain Natriuretic Peptide and troponin assessment | 7 months
  To correlate diastolic myocardial elasticity with a 6-minute walk test, Brain Natriuretic Peptide and troponin.

CONTACTS AND LOCATIONS:
Locations (1):
- Instituto do Coração - Hospital das Clínicas da Faculdade de Medicina da Universidade de São Paulo, São Paulo, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: No